CLINICAL TRIAL: NCT07024849
Title: Developing an Ecological and Tailored Nutritional Intervention to Improve Quality of Life in Esophageal Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Juhee Cho, Director of Cancer Education Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-05-127; RS-2023-CC139778 (Other Grant/Funding Number: Korean Cancer Survivor Healthcare R&D Project (National Cancer Center, funded by the Ministry of Health & Welfare))
Record Dates: First submitted 2025-05-12; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Cancer
Keywords: nutritional intervention; nutrition; survivors; esophageal cancer; care foods; health behavior; ecological intervention
MeSH Terms: conditions — Esophageal Neoplasms; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Intervention group (Experimental): This is a single-arm study, with all participants in the intervention arm. Patients in the intervention arm will receive a 4-week nutrition management program.
  Interventions: Dietary Supplement: Ecological nutritional intervention

INTERVENTIONS:
Dietary Supplement: Ecological nutritional intervention — Patients in the intervention arm will receive a 4-week nutrition management program(1 week for patients more than 4 months post-surgery), which includes providing nutritional guidelines, home delivery of personalized care foods, encouragement of physical activity using a wearable device, and weekly phone calls to check on nutritional goals and symptoms. Management services are also available through the mobile application.

SUMMARY:
This study aims to apply and assess the clinical feasibility of a health behavior theory-based ecological nutrition intervention program, providing nutrition care tailored to the unmet needs of esophageal cancer survivors after surgery.

Esophageal cancer survivors will receive a 4-week nutrition intervention program tailored to their individual nutritional needs. The program includes providing nutritional guidelines, customized care food, encouraging walking through a wearable device, and weekly telephone counseling. The evaluation of the program will assess food intake, adherence to dietary guidelines, activity level, nutritional indicators (such as PNI and NRI), weight change, fatigue, symptoms, quality of life, and satisfaction with meals and services. Additionally, interviews will be conducted after the intervention to evaluate the patient's experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical stage 1-3 primary esophageal cancer at diagnosis who have planned or received treatment, including esophageal resection and reconstruction, with curative intent, and their families*.
* You are at least 18 years of age
* Have a native-level understanding of Korean
* Who consented to this study

Exclusion Criteria:

* Concurrent multiple cancers at the time of diagnosis or a history of diagnosed and treated other organ cancers within the past year at the time of diagnosis
* Have had esophageal resection and reconstruction surgery for other reasons before being diagnosed with esophageal cancer
* Persons with limited cognitive and communication abilities
* The patient has had problems progressing to oral feeding after surgery, requiring a concurrent ileostomy, or the investigator determines that an interventional study is not appropriate.
* Individuals with reduced renal function for whom protein intake is not recommended (estimated GFR <60 mL/min/1.73 m2)
* People who are unable to walk due to joint problems, paralysis, etc.
* Those who do not use smartphones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Survey Questionnaire on Health Behavior Change through an Intervention Program | Baseline, end of intervention (post-enrollment 4 weeks)
  Adherence to nutritional guidelines including food intake

SECONDARY OUTCOMES:
Change in body weight (kg) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in body weight measured in kilograms from baseline to end of intervention.
Change in body composition (fat mass and fat-free mass) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in body composition assessed by bioimpedance analysis or DXA scan from baseline to end of intervention.
Change in Body Mass Index (BMI) (kg/m²) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in BMI calculated from weight and height from baseline to end of intervention.
Change in Patient-Generated Subjective Global Assessment Short Form (PG-SGA-SF) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in nutritional status assessed by the Patient-Generated Subjective Global Assessment Short Form (PG-SGA-SF) questionnaire (score range: 0-35, higher score indicates worse nutritional status) from baseline to end of intervention.
Change in Gastrointestinal Symptom Rating Scale (GSRS) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in gastrointestinal symptoms assessed by the Gastrointestinal Symptom Rating Scale (GSRS) questionnaire (score range: 1-7, higher score indicates more severe symptoms) from baseline to end of intervention.
Change in dumping syndrome assessed by clinical questionnaire | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in presence or severity of dumping syndrome assessed by clinical questionnaire or evaluation from baseline to end of intervention.
Change in EQ-5D-5L (EuroQol-5 Dimensions-5 Levels) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in quality of life assessed by the EQ-5D-5L questionnaire (score range: 0-1, higher score indicates better quality of life) from baseline to end of intervention.
Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in quality of life assessed by the EORTC QLQ-C30 (The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30) questionnaire (score range varies by domain; higher score in function scales indicates better function, higher score in symptom scales indicates worse symptoms) from baseline to end of intervention.
Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Oesophageal Cancer Module (EORTC QLQ-OES18) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in quality of life specific to esophageal cancer assessed by the EORTC QLQ-OES18 (The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Oesophagus 18) questionnaire (score range varies by domain; higher score in function scales indicates better function, higher score in symptom scales indicates worse symptoms) from baseline to end of intervention.
Change in patient satisfaction assessed by satisfaction survey | End of intervention (post-enrollment 4 weeks)
  Change in patient satisfaction assessed by satisfaction survey (score range: specify, e.g., 1-5, higher score indicates higher satisfaction) from baseline to end of intervention.
Service-experience assessed by qualitative interview | End of intervention (post-enrollment 4 weeks)
  Qualitative assessment of service experience through interview at end of intervention.

OTHER OUTCOMES:
Change in grip strength (kg) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in hand grip strength measured in kilograms from baseline to end of intervention.
Change in serum albumin (g/dL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in serum albumin level from baseline to end of intervention.
Change in prealbumin (mg/dL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in prealbumin level from baseline to end of intervention.
Change in Nutritional Risk Index (NRI) (score) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in Nutritional Risk Index score calculated from serum albumin and body weight from baseline to end of intervention.
Change in Prognostic Nutritional Index (PNI) score | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in Prognostic Nutritional Index score calculated from serum albumin and total lymphocyte count from baseline to end of intervention.
Change in total protein measured by laboratory assay (g/dL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in total protein level measured by laboratory assay from baseline to end of intervention.
Change in hemoglobin measured by laboratory assay (g/dL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in hemoglobin level measured by laboratory assay from baseline to end of intervention.
Change in white blood cell count (WBC) measured by laboratory assay (×10³/μL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in white blood cell count measured by laboratory assay from baseline to end of intervention.
Change in absolute lymphocyte count (ALC) measured by laboratory assay (×10³/μL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in absolute lymphocyte count measured by laboratory assay from baseline to end of intervention.
Change in absolute neutrophil count (ANC) measured by laboratory assay (×10³/μL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in absolute neutrophil count measured by laboratory assay from baseline to end of intervention.
Change in platelet count (PLT) measured by laboratory assay (×10³/μL) | Baseline, end of intervention (post-enrollment 4 weeks)
  Change in platelet count measured by laboratory assay from baseline to end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Juhee Cho, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No